CLINICAL TRIAL: NCT05084625
Title: PACED-Patient-centred Digital Support During Adjuvant Endocrine Breast Cancer Treatment
Brief Title: PACED-digitized Support During Adjuvant Endocrine Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Stockholm (Other Government)
Collaborators: ScientificMed Tech AB (Unknown); AstraZeneca (Industry); Novartis Sverige AB (Unknown); Bröstcancerförbundet (Unknown); Stockholm South General Hospital (Other); Capio St Gorans hospital (Unknown); Karolinska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-02902
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer; Treatment Adherence; Quality of Life; Treatment Side Effects
Keywords: Digital support
MeSH Terms: conditions — Breast Neoplasms; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A- access to digitized support, an app (Experimental): Patients in Arm A will have access to digitized support-an app for 12 months from baseline in addition to standard follow-up.
  Interventions: Other: Digitized support
- Arm B-standard follow-up (No Intervention): Patients in Arm B-will continue with standard follow-up from baseline and onwards

INTERVENTIONS:
Other: Digitized support — Access to information about the disease, treatment, side effects and self-care
  Arms: Arm A- access to digitized support, an app

SUMMARY:
The research team want to investigate whether digital support, an app under preventive hormonal breast cancer treatment can lead to less late side effects, better quality of life and increased adherence to treatment.

DETAILED DESCRIPTION:
Patients with hormon receptor positive breast cancer and adjuvant endocrine treatment will be invited to participate in the study after adjuvant radiotherapy is completed. Participants will be randomised to 12 months of access to a digital support-an app-in addition to standard follow-up or standard follow-up. Research team want to investigate whether digital support under hormonal breast cancer treatment can lead to less late side effects, better quality of life and increased adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Hormone receptor positive breast cancer
* On adjuvant endocrine treatment 0-16 weeks ago

Exclusion Criteria:

* Cognitively impaired
* No access to a mobile phone or internet
* Not understanding Swedish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Difference between the two groups with regard to change in quality of life from baseline to 12 months measured by Questionnaires European Organisation for Research and Treatment for Cancer Quality of life C30 (EORTC QLQ C30). | Change from baseline to 12 months
  EORTC QLQ C30. All of the scales and single-item measures range in score from 0 to100. A high scale score represents a higher response level. For a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems. A 'little' change for better or worse on a particular scale (function or symptom) defined as changes about 5 to 10. "Moderate" change have changed about 10 to 20, and 'very much' change corresponded to a change greater than 20. Our population sample is based on that a change should be of effect size (Cohen's d) difference of 0.54 (which correspond to a moderate change) at the end of access to digital support in the primary outcome of symptom burden and quality of life, 90% power at P < .01
Difference between the two groups with regard to change in quality of life from baseline to 12 months by Questionnaires European Organisation for Research and Treatment for Cancer Quality of life Breast cancerrelated 23 (EORTC QLQ BR23) | Change from baseline to 12 months
  EORTC QLQ BR23. All of the scales and single-item measures range in score from 0 to100. A high scale score represents a higher response level. For a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems. A 'little' change for better or worse on a particular scale (function or symptom) defined as changes about 5 to 10. "Moderate" change have changed about 10 to 20, and 'very much' change corresponded to a change greater than 20. BR23 recommended with C30. Our population sample is based on that a change should be of effect size (Cohen's d) difference of 0.54 (which correspond to a moderate change) at the end of access to digital support in the primary outcome of symptom burden and quality of life, 90% power at P < .01

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Bergqvist, Principal Investigator — St Gorans Hospital
Locations (3):
- Sweden (3):
  - Karolinska University Hospital, Stockholm
  - Oncology department Capio St Gorans Hospital, Stockholm
  - Södersjukhuset, Stockholm